CLINICAL TRIAL: NCT01781533
Title: An Open, Single-centre, Non-controlled Feasibility Study Using a Software-algorithm Based Insulin Therapy to Control Blood Glucose in Type 1 Diabetic Patients
Brief Title: Study to Test Software Algorithm for Insulin Therapy and New Glucose Sensor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Pieber Thomas, MD, Univ. Prof. Dr. med., Medical University of Graz
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: REACTbyALGO-1
Record Dates: First submitted 2013-01-23; First posted 2013-02-01 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Algorithms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- algorithm (Experimental)
  Interventions: Procedure: algorithm

INTERVENTIONS:
Procedure: algorithm

SUMMARY:
To investigate the performance of a software-algorithm based insulin therapy to control blood glucose in Type 1 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 to 75 years (both inclusive)
* Informed consent obtained after being advised of the nature of the study
* The subject has Type 1 diabetes (as defined by WHO) for at least 24 months
* The subject's HbA1c <= 10%
* Body Mass Index (BMI) <= 35 kg/m2
* The subject is treated with continuous subcutaneous insulin infusion for at least 3 month

Exclusion Criteria:

* Subject is actively enrolled in another clinical trial or took part in a study within 30 days
* Experienced recurrent severe hypoglycaemic unawareness
* Total daily insulin dose >= 1.4 IU/kg
* Subject is using a medication that significantly impacts glucose metabolism (oral or topical steroids) except if stable for at least the last three months and expected to remain stable for the study duration
* Allergy against insulin Lispro
* A history of drug or alcohol dependence
* Any other significant concomitant disease such as endocrine, cardiac, neurological, malignant, other pancreatic disease or uncontrolled hypertension as judged by the investigator
* Uncontrolled hypertension with resting blood pressure over 140/90 mmHg
* Patient is pregnant, or breast feeding during the period of the study
* Patient donated blood in the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
the percentage of glucose values obtained every 15 min in predefined glucose ranges | 15 minutes

SECONDARY OUTCOMES:
Injected insulin dose | 24 hours
Accuracy of the glucose monitoring unit | 24 hours
  The absolute and relative difference between glucose monitoring readings and reference values (blood glucose) will be used to determine the accuracy of the monitoring unit

CONTACTS AND LOCATIONS:
Overall Officials: Thomas R Pieber, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Styria, Austria